CLINICAL TRIAL: NCT05942872
Title: Immune Checkpoint Inhibitors Neurotoxicity: Long-term Outcomes, Predictors, and Survival.
Brief Title: CICLOPS Immune Checkpoint Inhibitors Neurotoxicity: Long-term Outcomes, Predictors, and Survival.
Acronym: LOPF - NIRAES
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 474
Record Dates: First submitted 2023-03-06; First posted 2023-07-12 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: Paraneoplastic Syndromes
Keywords: ICIs; NirAEs; paraneoplastic neurological syndromes; Neurological toxicity; immune checkpoint inhibitors
MeSH Terms: conditions — Paraneoplastic Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- NirAEs, grade ≥ 3 according to CTCAE: Patients treated with ICIs who developed neurologic syndromes consistent with NirAEs, of grade ≥ 3 according to the Common Terminology Criteria for Adverse Events (CTCAE)
  Interventions: Other: This is a non-interventional study. We will collect clinical data exclusively, and will do so by reviewing all available patients clinical records.

INTERVENTIONS:
Other: This is a non-interventional study. We will collect clinical data exclusively, and will do so by reviewing all available patients clinical records. — This is a non-interventional study. We will collect clinical data exclusively, and will do so by reviewing all available patients clinical records.

SUMMARY:
Immune-checkpoint inhibitors (ICIs) have radically changed the therapy of cancer in recent years. ICIs promote antitumor immune response inhibiting one of the following immune checkpoints: cytotoxic T-lymphocyte antigen-4 (CTLA-4; ipilimumab), programmed death-1 (PD-1: pembrolizumab, nivolumab, and cemiplimab), and programmed death ligand-1 (PD-L1: atezolizumab, durvalumab, and avelumab). Despite the desired effect as cancer treatment, ICIs can break immune tolerance to self-antigens and induce specific toxicities known as immune-related adverse events (irAEs), that may affect both peripheral and central nervous system (Neurological immune mediated adverse events, NirAEs). The pathogenic mechanisms underlying NirAEs are probably heterogeneous, as reflected by the variety of clinical phenotypes and severity.

NirAEs are rare, but there is some concern that the incidence may increase in the next future, in particular because ICIs are being used more and more for cancers commonly associated with paraneoplastic neurological syndromes (e.g. small-cell lung cancer). Moreover, NirAEs are usually severe, and often fatal. Indeed, irAEs-related complications are the most common cause of death among these patients. On the other hand, these patients usually have a good tumor response to immunotherapy. There is some evidence that irAEs may predict ICIs efficacy and consequently NirAE surivors are likely to have longer life expectancy than non-NirAE patients.

Therefore, it is of utmost importance to better characterize the long-term outcomes of NirAE patients in terms of neurologic disability and mortality, and to identify predictors of severe NirAEs. So far, only few studies with sufficient follow-up have been published on the topic, and they included only small number of patients.

The aims of our study is to characterize the main clinical and paraclinical features of NirAEs in a large cohort of NirAE patients, to assess long-term outcomes and to identify prognostic factors. This study will help define new guidelines regarding NirAE prediction and management.

ELIGIBILITY:
Inclusion Criteria:

* patients who developed NirAEs (grade severity equal or more than 3 according to CTCAE)

Exclusion Criteria:

* alternative better explanation for neurological symptoms (cancer progression, carcinomatous meningitis, complications of other treatments..)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with cancer treated with ICIs who experienced CTCAE grade ≥ 3 neurological toxicity (NirAEs)
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-07-15 (Actual); Study Completion 2021-09-15 (Actual)

PRIMARY OUTCOMES:
Prognostic factors in patients with NirAEs | Baseline (onset of NirAE) and 1 year.
  Evaluation of residual neurological disability as assessed by the modified Rankin scale (mRS)
  0 - No symptoms.
  1. - No significant disability. Able to carry out all usual activities, despite some symptoms.
  2. - Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.
  3. - Moderate disability. Requires some help, but able to walk unassisted.
  4. - Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.
  5. - Severe disability. Requires constant nursing care and attention, bedridden, incontinent.
  6. - Dead.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre de référence des syndromes neurologiques paranéoplasiques et encéphalites autoimmunes, Lyon, France